CLINICAL TRIAL: NCT00480714
Title: A Study of the Immunogenicity of M. Bovis BCG (SSI Strain), Delivered Intradermally in Healthy Volunteers
Brief Title: A Study of the Immunogenicity of BCG, Delivered Intradermally in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: TB003
Record Dates: First submitted 2007-05-30; First posted 2007-05-31 (Estimated); Last update posted 2007-05-31 (Estimated); Status verified 2007-05

CONDITIONS: TB
Keywords: TB; Vaccine; BCG

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: BCG (SSI Strain)

SUMMARY:
To assess the immunogenicity of M. bovis BCG (SSI strain), given intrademally in the standard dose used in clinical practice and to measure the development of the immune response in the first six months after administration. M. bovis BCG is a fully licensed vaccine that has been in routine clinical use for the last 50 years. It is the most widely administered vaccine in the world today and has an excellent safety record.

DETAILED DESCRIPTION:
Volunteers for the study will be recruited through advertisements. Each volunteer will have received an information sheet concerning the study and will have agreed to participate in writing.

Volunteers will be given at least 48 hours between reading the information leaflet and agreeing to participate. Female volunteers will have a pregnancy test prior to enrollment. Volunteers will give signed consent for their GP's to be notified about their participation in the trial. The GP will be faxed a letter on the day of screening and asked to reply if they know of a reason why the volunteer should not take part. The signed consent form will also be faxed with the letter.

A week after the screening visit and after a negative Heaf test, subjects will receive a single intradermal injection of 106 cfu M. bovis BCG in 0.1ml just inferior to the insertion of the deltoid muscle. Blood tests will be taken at the screening visit and day of immunisation, 1 and 2 weeks, and 1, 2, 3 and 6 months after the immunisation. 75mls will be taken on the screening visit, and 60mls will be taken on all subsequent visits. Screening samples will be tested for full blood count, biochemical screen and immunological assays to determine vaccine immunogenicity. Peripheral blood mononuclear cells will be prepared for cellular immunological assays to be performed without or following cryopreservation. Other serological measures of immune response, i.e.

antibody titres, will be assayed on frozen plasma samples. All blood tests will be taken within 1-3 days of the due date as described in the schedule above.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult aged 18-65 years.
* Normal medical history and physical examination.
* Normal urine dipstick, blood count, liver enzymes, and creatinine.

Exclusion Criteria:

* Exposure to TB/BCG vaccination at any point. Previous residence in a TB endemic area.
* Clinically significant history of skin disorder (eczema, psoriasis, etc.), allergy, immunodeficiency, cardiovascular disease, respiratory disease, endocrine disorder, liver disease, renal disease, gastrointestinal disease, neurological illness, psychiatric disorder, drug or alcohol abuse.
* Oral or systemic steroid medication or the use of immunosuppressive agents.
* Positive HIV or core HBV antibody test.
* Positive Heaf test
* Positive ANA or serum anti-DNA antibody.
* Confirmed pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2003-03; Study Completion 2003-09 (Actual)

PRIMARY OUTCOMES:
The induction of T-cell responses | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Helen I McShane, Principal Investigator — University of Oxford
Locations (1):
- University of Oxford, CCVTM, Churchill Hospital, Oxford, Oxfordshire, United Kingdom

REFERENCES:
- [Result] McShane H, Pathan AA, Sander CR, Keating SM, Gilbert SC, Huygen K, Fletcher HA, Hill AV. Recombinant modified vaccinia virus Ankara expressing antigen 85A boosts BCG-primed and naturally acquired antimycobacterial immunity in humans. Nat Med. 2004 Nov;10(11):1240-4. doi: 10.1038/nm1128. Epub 2004 Oct 24. PMID 15502839
- [Derived] Pathan AA, Sander CR, Fletcher HA, Poulton I, Alder NC, Beveridge NE, Whelan KT, Hill AV, McShane H. Boosting BCG with recombinant modified vaccinia ankara expressing antigen 85A: different boosting intervals and implications for efficacy trials. PLoS One. 2007 Oct 24;2(10):e1052. doi: 10.1371/journal.pone.0001052. PMID 17957238